CLINICAL TRIAL: NCT04939142
Title: A Phase III Randomized, Controlled, Multicenter, Open-label Study of ATG-010, Bortezomib, and Dexamethasone (SVd) Versus Bortezomib and Dexamethasone (Vd) in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of Evaluating the Safety and Efficacy of ATG-010, Bortezomib, and Dexamethasone (SVd) Versus Bortezomib and Dexamethasone (Vd) in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Acronym: BENCH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-MM-002
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SVd (Selinexor+Bortezomib+dexamethasone) (Experimental): Enrolled patients will be treated with ATG-010( 100 mg/QW, oral ) with Bortezomib( 1.3 mg/QW, hypodermic injection ) +dexamethasone ( 20 mg/QW, oral ) about 13.5cycles.
  Interventions: Combination Product: SVd (Selinexor+Bortezomib+dexamethasone)
- Vd(Bortezomib+dexamethasone) (Experimental): Enrolled patients will be treated with Bortezomib( 1.3 mg/QW, hypodermic injection ) +dexamethasone ( 20 mg/QW, oral ) about 13.5 cycles.
  Interventions: Combination Product: Vd (Bortezomib+dexamethasone)

INTERVENTIONS:
Combination Product: SVd (Selinexor+Bortezomib+dexamethasone) — Randomized into two treatment Arms in a 2:1 allocation (SVd Arm or Vd Arm): (1) SVd Arm (~100): ATG-010 + (Once a week, QW) + bortezomib (QW) + dexamethasone (BIW)
  Arms: SVd (Selinexor+Bortezomib+dexamethasone)
Combination Product: Vd (Bortezomib+dexamethasone) — Vd Arm (~50): Bortezomib (Cycles 1-8 [BIW], Cycles ≥ 9 [QW]) + dexamethasone (Cycles 1-8 [Four times a week], Cycles ≥ 9 [BIW])
  Arms: Vd(Bortezomib+dexamethasone)

SUMMARY:
This is a Phase III Randomized, Controlled, Multicenter, Open-label Study of ATG-010, Bortezomib, and Dexamethasone (SVd) Versus Bortezomib and Dexamethasone (Vd) in Patients with Relapsed or Refractory Multiple Myeloma (RRMM).

DETAILED DESCRIPTION:
This is a Phase III Randomized, Controlled, Multicenter, Open-label Study of ATG-010, Bortezomib, and Dexamethasone (SVd) Versus Bortezomib and Dexamethasone (Vd) in Patients with Relapsed or Refractory Multiple Myeloma (RRMM). About 150 subjects are planned to be enrolled in this study, and be randomized into two treatment Arms in a 2:1 allocation (SVd Arm or Vd Arm).

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form (ICF).
2. Age ≥ 18 years.
3. Confirmed MM with measurable disease per IMWG guidelines, and meet at least 1 of the following:

   1. Serum M-protein ≥ 0.5 g/dL (> 5 g/L) by serum protein electrophoresis (SPEP) or for immunoglobulin IgA, IgD myeloma, replaced by quantitative serum IgA, IgD levels; or
   2. Urinary M-protein level ≥ 200 mg/24 hours; or
   3. Serum FLC ≥ 100 mg/L, provided that the serum FLC ratio is abnormal (Normal FLC ratio: 0.26 to 1.65).
4. Had at least 1 prior anti-MM regimen and no more than 3 prior anti-MM regimens. Induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 anti-MM regimen.
5. Valid evidence of progressive MM (based on the Investigator's determination according to the IMWG response criteria) on or after their last regimen.
6. Must have an ECOG Status score of 0, 1, or 2.
7. Renal function should meet the following criteria: creatinine clearance [CrCl] rates ≥ 20 mL/min (Calculated using the formula of Cockroft and Gault).
8. Resolution of any clinically significant non-hematological toxicities (If any) from previous treatments to Grade ≤1 or baseline by C1D1. Subject with chronic, stable Grade 2 non hematological toxicities may be included following approval from the Medical Monitor.
9. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening. Female subjects of childbearing potential and fertile male subjects must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

1. Prior exposure to SINE compounds (Including ATG-010), or suspected allergy to SINE or similar drugs.
2. Active plasma cell leukemia.
3. Documented systemic light chain amyloidosis.
4. MM involving the central nervous system.
5. POEMS syndrome (Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes).
6. Spinal cord compression related to MM.
7. Greater than Grade 2 peripheral neuropathy or Grade ≥ 2 peripheral neuropathy with pain at baseline, regardless of whether the subject is currently receiving medication.
8. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
9. Active graft versus host disease (After allogeneic stem cell transplantation) at screening.
10. Uncontrolled active infections requiring intravenous antibiotics, antivirals, or antifungal therapy in 2 weeks prior to C1D1.
11. Major surgery within 4 weeks prior to C1D1.
12. Known active human immunodeficiency virus (HIV) infection or HIV seropositivity.
13. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus ribonucleic acid (RNA) or hepatitis B virus deoxyribonucleic acid (HBV-DNA).
14. Pregnant or lactating women.
15. Life expectancy of < 4 months.
16. Any active gastrointestinal dysfunction interfering with the subject's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
17. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
18. Contraindication to any of the required concomitant drugs or supportive treatments.
19. Any diseases or complications which may interfere with the study procedures.
20. Subject unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Three years after last patient first dose
  To evaluate progression-free survival

SECONDARY OUTCOMES:
Overall Survival (OS) | Three years after last patient first dose
  The estimates of Kaplan-Meier
Duration of Response (DOR) | Three years after last patient first dose
  To evaluate duration of response
Objective response rate (ORR) | Three years after last patient first dose
  evaluated by IRC (PR + VGPR + CR + sCR)
Progression-free survival(PFS2) | Three years after last patient first dose
  PFS after further treatment followed by treatment with SVd/Vd
Time to remission(TTR) | Three years after last patient first dose
  To compare the efficacy of treatment with SVd and Vd
VGPR+CR+sCR | Three years after last patient first dose
  Proportion of subjects of VGPR + CR + sCR
Safety Endpoints | Three years after last patient first dose
  Incidence of any Grade ≥ 2 peripheral neuropathy events

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, PhD, Principal Investigator — Peking University People's Hospital
Locations (33):
- China (33):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital OF USTC, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital Army Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People'S Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Shenzhen Second People'S Hospital, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Nantong University, Nanchang, Jiangxi
  - The First Hospital of Nanchang, Nanchang, Jiangxi
  - Shengjing Hospital China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Qilu Hospital of Shangdong University, Jinan, Shangdong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital Zhejiang University of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang